CLINICAL TRIAL: NCT06343402
Title: A Phase 1a/1b Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of BBO-8520 in Subjects With Advanced KRASG12C Mutant Non-Small Cell Lung Cancer - The ONKORAS-101 Study
Brief Title: Open-label Study of BBO-8520 in Adult Subjects With KRASG12C Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TheRas, Inc., d/b/a BBOT (BridgeBio Oncology Therapeutics) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TBBO8520-101; ONKORAS-101 (Other: TheRas, Inc., d/b/a BBOT (BridgeBio Oncology Therapeutics))
Record Dates: First submitted 2024-03-22; First posted 2024-04-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer; Metastatic Non-Small Cell Lung Cancer; NSCLC; KRAS G12C; Metastatic Lung Cancer; Advanced Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1a: sequential/parallel, Phase 1b: parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1a - Dose Escalation/Dose Finding Monotherapy (Experimental): Participants enrolled in this cohort will receive BBO-8520 (different dose levels will be evaluated) once a day (QD) as monotherapy
  Interventions: Drug: BBO-8520
- Cohort 1b - Dose Escalation/Dose Finding Combination Therapy (Experimental): Participants enrolled in this cohort will receive BBO-8520 (different dose levels will be evaluated) once a day (QD) in combination with pembrolizumab infusion (IV)
  Interventions: Drug: BBO-8520; Drug: Pembrolizumab
- Cohort 2a - Dose Expansion Monotherapy (Experimental): Participants enrolled in this cohort will receive BBO-8520 once a day (QD) as monotherapy
  Interventions: Drug: BBO-8520
- Cohort 2b - Dose Expansion Combination Therapy (Experimental): Participants enrolled in this cohort will receive BBO-8520 once a day (QD) in combination with pembrolizumab infusion (IV)
  Interventions: Drug: BBO-8520; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BBO-8520 — Participants will receive assigned dose of BBO-8520 orally (PO), QD
Drug: Pembrolizumab — Patients will receive IV pembrolizumab
  Arms: Cohort 1b - Dose Escalation/Dose Finding Combination Therapy; Cohort 2b - Dose Expansion Combination Therapy

SUMMARY:
A first in human study to evaluate the safety and preliminary antitumor activity of BBO-8520, a KRAS G12C (ON and OFF) inhibitor, as a single agent and in combination with pembrolizumab in subjects with locally advanced and unresectable or metastatic non-small cell lung cancer with a KRAS (Kirsten rat sarcoma) G12C mutation.

DETAILED DESCRIPTION:
This is an open-label, multi-center, Phase 1 study designed to evaluate the safety, tolerability, pharmacokinetics, and efficacy of BBO-8520, a direct inhibitor of KRASG12C (ON and OFF), alone and in combination with the ICI pembrolizumab in subjects with locally advanced and unresectable or metastatic non-small cell lung cancer with a KRAS (Kirsten rat sarcoma) G12C mutation. The study includes dose escalation phase and dose expansion phase

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented locally advanced and unresectable or metastatic non-small cell lung cancer with a KRAS G12C mutation
* Measurable disease by RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1

Exclusion Criteria:

* Patients with malignancy within the last 2 years as specified in the protocol
* Patients with untreated brain metastases
* Patients with known hypersensitivity to BBO-8520 or its excipients
* For Cohorts 1b and 2b:
* Patients with a known hypersensitivity to pembrolizumab or its excipients
* Patients with active autoimmune disease of history of autoimmune disease that might recur
* Patients with a history of interstitial lung disease/pneumonitis that required steroids, or current interstitial lung disease/pneumonitis

Other inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | approximately 3 years
  Incidence and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs)
Dose-limiting toxicities (DLTs) | approximately 3 years
  Number of participants with dose limiting toxicities

SECONDARY OUTCOMES:
To evaluate preliminary antitumor activity of BBO-8520 | approximately 3 years
  Objective response rate (ORR) per (RECIST v1.1)
To evaluate preliminary antitumor activity of BBO-8520 | approximately 3 years
  Duration of Response (DOR) per (RECIST v1.1)
To evaluate preliminary antitumor activity of BBO-8520 | approximately 3 years
  Progression-free survival (PFS) per (RECIST v1.1)
Overall Survival (OS) | approximately 3 years
To characterize the pharmacokinetics (PK) of BBO-8520 | approximately 3 years
  Area under the curve (AUC)
To characterize the pharmacokinetics (PK) of BBO-8520 | approximately 3 years
  Peak plasma drug concentration (Cmax)
To characterize the pharmacokinetics (PK) of BBO-8520 | approximately 3 years
  Time to Cmax (Tmax)
To characterize the pharmacokinetics (PK) of BBO-8520 | approximately 3 years
  Half life (T1/2)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (18):
  - University of California - San Diego Moores Cancer Center, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - UCLA Health - Santa Monica Cancer Care, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry Ford Cancer - Detroit, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Perlmutter Cancer Center - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - Oncology Consultants Texas Medical Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - NEXT Oncology, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Northwest Medical Specialties, Tacoma, Washington
- Australia (6):
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Peninsula & South Eastern Hematology and Oncology Group (PAS), Frankston, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Canada (3):
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec